CLINICAL TRIAL: NCT01445301
Title: Study STF115287, a Clinical Confirmation Study of GSK2585823 (Clindamycin 1%-Benzoyl Peroxide 3% Gel) in the Treatment of Acne Vulgaris in Japanese Subjects. - A Multicenter, Randomized, Single-blind, Active-controlled, Parallel-group Study -
Brief Title: Study STF115287, a Clinical Confirmation Study of GSK2585823 in the Treatment of Acne Vulgaris in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 115287
Record Dates: First submitted 2011-09-15; First posted 2011-10-03 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2017-09

CONDITIONS: Acne Vulgaris
Keywords: twice daily; once daily; CLDM 1%-BPO 3% gel; Clindamycin (CLDM); benzoyl peroxide (BPO); inflammatory lesion; non-inflammatory lesion; acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GSK2585823(CLDM 1%-BPO 3% gel) once daily (Experimental): Subjects will apply in a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin). Also, the dose regimen will be once daily in the evening/bedtime.
  Interventions: Drug: GSK2585823(CLDM 1%-BPO 3% gel)
- GSK2585823(CLDM 1%-BPO 3% gel) twice daily (Experimental): Subjects will apply in a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin). Also, the dose regimen will be twice daily in the morning and evening/bedtime.
  Interventions: Drug: GSK2585823(CLDM 1%-BPO 3% gel)
- CLDM 1% gel twice daily (Active Comparator): Subjects will apply in a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin). Also, the dose regimen will be twice daily in the morning and evening/bedtime.
  Interventions: Drug: CLDM 1% gel twice daily

INTERVENTIONS:
Drug: GSK2585823(CLDM 1%-BPO 3% gel) — Topical gel in 1 g containing clindamycin 10 mg and benzoyl peroxide 30 mg
  Other Names: GSK2585823
  Arms: GSK2585823(CLDM 1%-BPO 3% gel) once daily; GSK2585823(CLDM 1%-BPO 3% gel) twice daily
Drug: CLDM 1% gel twice daily — Topical gel containing clindamycin 10 mg/1 g gel
  Other Names: CLDM
  Arms: CLDM 1% gel twice daily

SUMMARY:
This is a multicenter, randomized, single-blinded (investigator's blinded), active-controlled (clindamycin [CLDM] 1% gel), parallel-group study in Japanese subjects with acne vulgaris to demonstrate the efficacy of GSK2585823 (CLDM 1%-benzoyl peroxide [BPO] 3% gel) when applied once or twice daily for 12 weeks. This study will also evaluate the safety of GSK2585823 when applied topically either once or twice daily for 12 weeks.

DETAILED DESCRIPTION:
Main inclusion criteria will be 12 to 45 years of age, who have an Investigator Static Global Assessment (ISGA) score of 2 or greater at baseline visit, and have both 17 to 60 facial inflammatory lesions (papules plus pustules) and 20 to 150 facial non-inflammatory lesions (open and closed comedones), including nasal lesions. The primary objectives are to demonstrate the superiority of GSK2585823 twice daily to CLDM twice daily in total lesion counts, and to demonstrate the non-inferiority of GSK2585823 once daily to CLDM twice daily in total lesion counts. The secondary objectives are to demonstrate the non-inferiority of GSK2585823 once daily to CLDM twice daily in inflammatory lesion counts, and to evaluate the efficacy of GSK2585823 once or twice daily compared with CLDM twice daily at each visit. A total of 800 subjects will be enrolled and randomly assigned to one of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 12 to 45 years (inclusive) of age in good general health.
* Subjects must have both on the face:

A) A minimum of 17 but not more than 60 inflammatory lesions (papules/pustules), including nasal lesions.

And B) A minimum of 20 but not more than 150 non-inflammatory lesions (open/closed comedones), including nasal lesions.

* An ISGA score of 2 or greater at baseline.
* Females of childbearing potential and women who are less than 2 years from their last menses must agree to use the contraception.
* The ability and willingness to follow all study procedures and attend all scheduled visits.
* The ability to understand and sign a written informed consent form (Written informed consent must be obtained also from the parent or guardian in case of subject under 20 years of age at the time of given consent).

Exclusion Criteria:

* Have any nodule-cystic lesions at baseline.
* Are pregnant or breast-feeding.
* Have a history or presence of regional enteritis, inflammatory bowel disease (e.g., ulcerative colitis, pseudomembranous colitis, chronic diarrhea or antibiotic-associated colitis) or similar symptoms.
* Used any of the following agents on the face within the previous 2 weeks:Topical antibiotics (or systemic antibiotics);Topical anti-acne medications (e.g., BPO, azelaic acid, resorcinol, salicylates);Abradants, facials, or peels containing glycolic or other acids;Masks, washes or soaps containing BPO, sulfacetamide sodium, or salicylic acid;Non-mild facial cleansers (e.g., facial scrub, cleansers containing agents with anti-inflammatory action); Moisturizers that contain retinol, salicylic acid, or α- or β-hydroxy acids;Astringents and toner (Subjects are allowed to enroll in this study, if the subject has been on treatment for more than 2 consecutive weeks prior to start of investigational product use).
* Used the following agents on the face or performed the following procedure within the previous 4 weeks:Topical corticosteroids (Use of inhaled, intra-articular, or intra-lesional steroids other than for facial acne is acceptable);Facial procedure (such as chemical or laser peel, microdermabrasion, blue light treatment, etc.).
* Used systemic retinoids within the previous 6 months or topical retinoids on the face within the previous 6 weeks.
* Received treatment with estrogens, androgens, or anti-androgenic agents within the previous 12 weeks (Subjects who have been treated with the above agents for more than 12 consecutive weeks prior to start of investigational product are allowed to enrol as long as they do not expect to change dose, drug, or discontinue use during the study).
* Used any medication that in the opinion of the investigator may affect this clinical study or evaluation of the study.
* Plan to use medications that are reported to exacerbate acne (e.g., mega-doses of certain vitamins, such as vitamin D [>2000 IU/day] and vitamin B12 [>1 mg/day], corticosteroids*, androgens, haloperidol, halogens [e.g., iodide and bromide], lithium, hydantoin, and phenobarbital).

  *: except the using of topical corticosteroids (e.g., inhaled, intra-articular, or intra-lesional steroids) other than for facial acne.
* Have a known hypersensitivity or have had previous allergic reaction to any of the components of the investigational product.
* Used any investigational therapy within the previous 12 weeks, or plan to participate in another clinical study at the same time.
* Participated in Japanese clinical studies planned by GlaxoSmithKline K.K. in the development of investigational products for acne vulgaris.
* Are currently abusing drugs or alcohol.
* Have a significant medical history of being immunocompromised.
* People as follows and the family members:Employees of GlaxoSmithKline, contract research organization (CRO) or site management organization (SMO);Investigators.
* Have other conditions that would put the subject at unacceptable risk for participation in the study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Actual)
Dates: Start 2011-09-27 (Actual); Primary Completion 2012-08-02 (Actual); Study Completion 2012-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Japan (6):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 800 Japanese participants across 26 investigational centers in Japan, with Acne Vulgaris were enrolled in this study. The study was conducted from 27 September 2011 - 02 August 2012.
Groups:
- GSK2585823 Once Daily: Participants were instructed to apply GSK2585823 (Topical gel in 1 gram (g) containing clindamycin (CLDM) 10 milligram (mg) and benzoyl peroxide 30 mg) a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin) once daily in the evening/bedtime for 12 weeks. The indication of application volume was 2 FTU (Finger Tip Unit).
- GSK2585823 Twice Daily: Participants were instructed to apply GSK2585823 (Topical gel in 1 g containing CLDM 10 mg and benzoyl peroxide 30 mg) a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin) twice daily in the morning and evening/bedtime for 12 weeks. The indication of application volume was 2 FTU.
- CLDM Twice Daily: Participants were instructed to apply CLDM (topical gel containing CLDM 10 mg/1 g gel) that is Dalacin® T Gel 1% a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin) twice daily in the morning and evening/bedtime for 12 weeks. The indication of application volume was 2 FTU.
Period: Overall Study
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Started | 204 | 297 | 299
Completed | 183 | 262 | 290
Not Completed | 21 | 35 | 9
Not completed — Adverse Event | 15 | 25 | 4
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Protocol-Defined Stopping Criteria | 0 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population comprised all randomized participants who received at least one application of investigational product. One participant excluded was randomized but was not administered study drug. 799 participant were included in the ITT population.
Groups:
- GSK2585823 Once Daily: Participants were instructed to apply GSK2585823 (Topical gel in 1 g containing CLDM 10 mg and benzoyl peroxide 30 mg) a quantity sufficient to cover the entire face (including the forehead, nose, cheeks, and chin) once daily in the evening/bedtime for 12 weeks. The indication of application volume was 2 FTU.
- Total: Total of all reporting groups
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily | Total
Number analyzed (Participants) | 204 | 296 | 299 | 799
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.4 (6.06) | 20.7 (6.33) | 21.1 (6.55) | 20.8 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 187 | 202 | 528
  Male | 65 | 109 | 97 | 271
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 204 | 296 | 299 | 799
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Week 12 in Total Lesion Counts.
Description: The investigator (or subinvestigator) counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedones) on the face at each study visit. An open comedone was an open, widely dilated follicle with black-colored sebum, due to melanin and oxidation, and keratinous material that forms a plug, thereby obstructing the pilosebaceous duct. A closed comedone was a closed follicle filled with impacted sebum covered by keratin that has a whitish color. A papule was a small, raised, red, dome-shaped palpable lesion. A pustule was a raised, dome-shaped palpable lesion containing yellow fluid (pus). A nodule might be a raised or deep-seated, dome-shaped palpable lesion of at least 5 millimeters in diameter. Day 1 was Baseline and change from baseline was calculated by subtracting the Baseline value from post-randomization value at Week 12.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 201 | 289 | 299
lesion count | -57.2 (1.94) | -60.8 (1.53) | -49.8 (1.52)
Statistical Analysis 1: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -11.0, 95% CI 2-sided [-15.0 to -7.0]
Statistical Analysis 2: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Test type: Non-Inferiority — If the upper 95% confidence was less than the pre-defined threshold (-Δ [non-inferiority margin, -3.8]) of 3.8, non-inferiority of GSK2585823 once daily to CLDM twice daily would be established; p < 0.001, ANCOVA; Mean Difference (Net) = -8.2, 95% CI 2-sided [-12.9 to -3.6]

2. Secondary Outcome: Absolute Change From Baseline to Weeks 1, 2, 4, and 8 in Total Lesion Counts
Description: The investigator (or subinvestigator) counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedones) on the face at each study visit. An open comedone was an open, widely dilated follicle with black-colored sebum, due to melanin and oxidation, and keratinous material that forms a plug, thereby obstructing the pilosebaceous duct. A closed comedone was a closed follicle filled with impacted sebum covered by keratin that has a whitish color. A papule was a small, raised, red, dome-shaped palpable lesion. A pustule was a raised, dome-shaped palpable lesion containing yellow fluid (pus). A nodule might be a raised or deep-seated, dome-shaped palpable lesion of at least 5 millimeters in diameter. Day 1 was Baseline and change from baseline was calculated by subtracting the Baseline value from value at indicated time points.
Time Frame: Baseline (Day 1) and Weeks 1, 2, 4, and 8
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
lesion count
  WEEK 1: number analyzed (Participants) | 200 | 287 | 295
  WEEK 1 | -22.9 (19.81) | -25.6 (24.91) | -16.9 (24.40)
  WEEK 2: number analyzed (Participants) | 201 | 289 | 299
  WEEK 2 | -32.9 (29.18) | -37.9 (28.91) | -26.6 (30.00)
  WEEK 4: number analyzed (Participants) | 201 | 289 | 299
  WEEK 4 | -41.4 (27.41) | -47.3 (31.04) | -34.8 (30.92)
  WEEK 8: number analyzed (Participants) | 201 | 289 | 299
  WEEK 8 | -49.1 (28.97) | -54.4 (34.65) | -42.7 (33.49)

3. Secondary Outcome: Absolute Change From Baseline to Weeks 1, 2, 4, 8, and 12 in Inflammatory and Non-inflammatory Lesion Counts
Description: as for outcome 2
Time Frame: Baseline (Day 1) and Weeks 1, 2, 4, 8, and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Lesion count
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
Lesion count
  Inflammatory lesions,Week 1: number analyzed (Participants) | 200 | 287 | 295
  Inflammatory lesions,Week 1 | -11.5 (0.60) | -11.1 (0.54) | -8.5 (0.50)
  Inflammatory lesions,Week 2: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions,Week 2 | -14.8 (0.90) | -16.4 (0.61) | -13.1 (0.76)
  Inflammatory lesions,Week 4: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions,Week 4 | -18.3 (0.93) | -19.1 (0.62) | -16.3 (0.78)
  Inflammatory lesions,Week 8: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions,Week 8 | -21.0 (0.98) | -21.3 (0.69) | -18.3 (0.82)
  Inflammatory lesions,Week 12: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions,Week 12 | -22.9 (0.99) | -23.3 (0.69) | -20.3 (0.83)
  Non-Inflammatory lesions,Week 1: number analyzed (Participants) | 200 | 287 | 295
  Non-Inflammatory lesions,Week 1 | -13.1 (1.26) | -15.6 (1.08) | -9.7 (1.06)
  Non-Inflammatory lesions,Week 2: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions,Week 2 | -20.3 (1.53) | -22.8 (1.28) | -14.9 (1.29)
  Non-Inflammatory lesions,Week 4: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions,Week 4 | -25.2 (1.58) | -28.9 (1.33) | -19.4 (1.32)
  Non-Inflammatory lesions,Week 8: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions,Week 8 | -30.4 (1.62) | -33.9 (1.36) | -24.9 (1.36)
  Non-Inflammatory lesions,Week 12: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions,Week 12 | -34.3 (1.60) | -37.5 (1.31) | -28.7 (1.34)
Statistical Analysis 1: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -3.0, 95% CI 2-sided [-4.4 to -1.5]
Statistical Analysis 2: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 2; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.113, ANCOVA; Mean Difference (Net) = -1.8, 95% CI 2-sided [-4.0 to 0.4]
Statistical Analysis 3: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.084, ANCOVA; Mean Difference (Net) = -2.0, 95% CI 2-sided [-4.2 to 0.3]
Statistical Analysis 4: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 8; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.026, ANCOVA; Mean Difference (Net) = -2.7, 95% CI 2-sided [-5.1 to -0.3]
Statistical Analysis 5: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 12; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.030, ANCOVA; Mean Difference (Net) = -2.6, 95% CI 2-sided [-5.0 to -0.3]
Statistical Analysis 6: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.028, ANCOVA; Mean Difference (Net) = -3.4, 95% CI 2-sided [-6.5 to -0.4]
Statistical Analysis 7: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 2; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.004, ANCOVA; Mean Difference (Net) = -5.4, 95% CI 2-sided [-9.1 to -1.7]
Statistical Analysis 8: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.003, ANCOVA; Odds Ratio (OR) = -5.8, 95% CI 2-sided [-9.6 to -1.9]
Statistical Analysis 9: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 8; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.006, ANCOVA; Mean Difference (Net) = -5.5, 95% CI 2-sided [-9.4 to -1.6]
Statistical Analysis 10: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; WEEK 12; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.005, ANCOVA; Mean Difference (Net) = -5.6, 95% CI 2-sided [-9.5 to -1.7]
Statistical Analysis 11: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 1; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -2.5, 95% CI 2-sided [-3.9 to -1.1]
Statistical Analysis 12: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 2; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -3.2, 95% CI 2-sided [-4.7 to -1.6]
Statistical Analysis 13: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 4; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = -2.5, 95% CI 2-sided [-4.1 to -0.9]
Statistical Analysis 14: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 8; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Net) = -2.7, 95% CI 2-sided [-4.5 to -0.9]
Statistical Analysis 15: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 12; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = -2.8, 95% CI 2-sided [-4.6 to -1.0]
Statistical Analysis 16: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 1; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -6.0, 95% CI 2-sided [-8.8 to -3.2]
Statistical Analysis 17: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 2; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -8.1, 95% CI 2-sided [-11.4 to -4.7]
Statistical Analysis 18: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 4; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -9.7, 95% CI 2-sided [-13.1 to -6.2]
Statistical Analysis 19: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 8; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -8.6, 95% CI 2-sided [-12.1 to -5.1]
Statistical Analysis 20: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; WEEK 12; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -8.2, 95% CI 2-sided [-11.6 to -4.8]

4. Secondary Outcome: Percent Change From Baseline to Weeks 1, 2, 4, 8, and 12 in Total, Inflammatory, and Non- Inflammatory Lesion Counts
Description: The investigator (or subinvestigator) counted all inflammatory lesions (papules, pustules, and nodular lesions) and non-inflammatory lesions (open and closed comedones) on the face at each study visit. An open comedone was an open, widely dilated follicle with black-colored sebum, due to melanin and oxidation, and keratinous material that forms a plug, thereby obstructing the pilosebaceous duct. A closed comedone was a closed follicle filled with impacted sebum covered by keratin that has a whitish color. A papule was a small, raised, red, dome-shaped palpable lesion. A pustule was a raised, dome-shaped palpable lesion containing yellow fluid (pus). A nodule might be a raised or deep-seated, dome-shaped palpable lesion of at least 5 millimeters in diameter. Day 1 was Baseline and change from baseline was calculated by subtracting the Baseline value from value at indicated time points.( Weeks 1, 2, 4, 8 and 12)
Time Frame: Baseline (Day 1) and Weeks 1, 2, 4, 8, and 12
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
Percent change
  Total lesions,Week 1: number analyzed (Participants) | 200 | 287 | 295
  Total lesions,Week 1 | -32.42 (1.478) | -33.29 (1.312) | -24.71 (1.247)
  Total lesions,Week 2: number analyzed (Participants) | 201 | 289 | 299
  Total lesions,Week 2 | -46.87 (1.953) | -49.29 (1.544) | -38.36 (1.644)
  Total lesions,Week 4: number analyzed (Participants) | 201 | 289 | 299
  Total lesions,Week 4 | -57.15 (1.848) | -59.98 (1.454) | -48.26 (1.556)
  Total lesions,Week 8: number analyzed (Participants) | 201 | 289 | 299
  Total lesions,Week 8 | -66.33 (1.935) | -68.49 (1.551) | -57.20 (1.630)
  Total lesions,Week 12: number analyzed (Participants) | 201 | 289 | 299
  Total lesions,Week 12 | -73.85 (1.929) | -75.57 (1.512) | -64.42 (1.625)
  Inflammatory lesions, Week 1: number analyzed (Participants) | 200 | 287 | 295
  Inflammatory lesions, Week 1 | -41.87 (1.885) | -39.76 (1.704) | -31.32 (1.590)
  Inflammatory lesions, Week 2: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions, Week 2 | -55.64 (2.277) | -58.31 (1.641) | -48.43 (1.917)
  Inflammatory lesions, Week 4: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions, Week 4 | -66.51 (2.181) | -66.89 (1.617) | -58.87 (1.837)
  Inflammatory lesions, Week 8: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions, Week 8 | -74.86 (2.256) | -74.37 (1.750) | -66.13 (1.899)
  Inflammatory lesions, Week 12: number analyzed (Participants) | 201 | 289 | 299
  Inflammatory lesions, Week 12 | -80.84 (2.120) | -81.14 (1.598) | -72.64 (1.785)
  Non-Inflammatory lesions, Week 1: number analyzed (Participants) | 200 | 287 | 295
  Non-Inflammatory lesions, Week 1 | -26.49 (1.846) | -29.20 (1.697) | -20.69 (1.558)
  Non-Inflammatory lesions, Week 2: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions, Week 2 | -41.26 (2.392) | -43.43 (2.022) | -32.96 (2.014)
  Non-Inflammatory lesions, Week 4: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions, Week 4 | -51.12 (2.246) | -55.40 (1.847) | -41.85 (1.891)
  Non-Inflammatory lesions, Week 8: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions, Week 8 | -60.59 (2.247) | -64.83 (1.844) | -51.75 (1.892)
  Non-Inflammatory lesions, Week 12: number analyzed (Participants) | 201 | 289 | 299
  Non-Inflammatory lesions, Week 12 | -69.01 (2.219) | -71.90 (1.804) | -59.33 (1.869)
Statistical Analysis 1: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -7.71, 95% CI 2-sided [-11.30 to -4.12]
Statistical Analysis 2: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -8.51, 95% CI 2-sided [-13.24 to -3.77]
Statistical Analysis 3: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -8.89, 95% CI 2-sided [-13.37 to -4.41]
Statistical Analysis 4: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 8; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -9.12, 95% CI 2-sided [-13.82 to -4.43]
Statistical Analysis 5: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 12; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -9.43, 95% CI 2-sided [-14.11 to -4.75]
Statistical Analysis 6: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -10.54, 95% CI 2-sided [-15.12 to -5.97]
Statistical Analysis 7: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.011, ANCOVA; Mean Difference (Net) = -7.21, 95% CI 2-sided [-12.73 to -1.69]
Statistical Analysis 8: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.005, ANCOVA; Mean Difference (Net) = -7.64, 95% CI 2-sided [-12.93 to -2.35]
Statistical Analysis 9: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 8; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.002, ANCOVA; Mean Difference (Net) = -8.73, 95% CI 2-sided [-14.20 to -3.26]
Statistical Analysis 10: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 12; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.002, ANCOVA; Mean Difference (Net) = -8.20, 95% CI 2-sided [-13.34 to -3.06]
Statistical Analysis 11: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.011, ANCOVA; Mean Difference (Net) = -5.80, 95% CI 2-sided [-10.29 to -1.32]
Statistical Analysis 12: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.005, ANCOVA; Mean Difference (Net) = -8.30, 95% CI 2-sided [-14.10 to -2.50]
Statistical Analysis 13: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -9.27, 95% CI 2-sided [-14.72 to -3.83]
Statistical Analysis 14: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 8; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.002, ANCOVA; Mean Difference (Net) = -8.84, 95% CI 2-sided [-14.28 to -3.39]
Statistical Analysis 15: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 12; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANCOVA; Mean Difference (Net) = -9.68, 95% CI 2-sided [-15.06 to -4.30]
Statistical Analysis 16: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 1; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -8.90, 95% CI 2-sided [-12.32 to -5.48]
Statistical Analysis 17: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 2; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -11.17, 95% CI 2-sided [-15.18 to -7.16]
Statistical Analysis 18: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 4; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -12.12, 95% CI 2-sided [-15.90 to -8.35]
Statistical Analysis 19: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 8; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -11.33, 95% CI 2-sided [-15.37 to -7.30]
Statistical Analysis 20: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Total Lesion Counts, WEEK 12; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -11.18, 95% CI 2-sided [-15.11 to -7.25]
Statistical Analysis 21: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 1; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -8.32, 95% CI 2-sided [-12.76 to -3.88]
Statistical Analysis 22: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 2; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -9.57, 95% CI 2-sided [-13.83 to -5.30]
Statistical Analysis 23: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 4; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -7.83, 95% CI 2-sided [-12.03 to -3.62]
Statistical Analysis 24: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 8; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -8.08, 95% CI 2-sided [-12.63 to -3.53]
Statistical Analysis 25: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Inflammatory Lesion Counts, WEEK 12; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -8.56, 95% CI 2-sided [-12.71 to -4.41]
Statistical Analysis 26: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 1; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -9.11, 95% CI 2-sided [-13.53 to -4.68]
Statistical Analysis 27: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 2; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -11.05, 95% CI 2-sided [-16.30 to -5.80]
Statistical Analysis 28: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 4; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -14.17, 95% CI 2-sided [-18.97 to -9.37]
Statistical Analysis 29: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 8; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -13.04, 95% CI 2-sided [-17.83 to -8.25]
Statistical Analysis 30: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Non-Inflammatory Lesion Counts, WEEK 12; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -12.37, 95% CI 2-sided [-17.05 to -7.68]

5. Secondary Outcome: Percentage of Participants With a Minimum 2-grade Improvement From Baseline to Week 12 in Investigator's Static Global Assessment (ISGA) Score
Description: Proportion of participants with at least a 2-Grade Improvement in ISGA was reported using a 5 point scale which indicates Score 0 (Clear): skin with no inflammatory or non-inflammatory lesions, Score 1 (Almost Clear): rare non-inflammatory lesions with no more than rare papules, Score 2 (Mild): greater than Grade 1, some non-inflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions), Score 3 (Moderate): greater than Grade 2, many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion, Score 4 (Severe): greater than Grade 3, many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions and 5(very severe): many non-inflammatory and inflammatory lesions and more than a few nodular lesions. May have cystic lesions. The investigator assessed ISGA score at baseline (Week 0/Day 1) and Weeks 1, 2, 4, 8, and 12. The area evaluated ISGA was limited to the face.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 184 | 262 | 290
Percentage of Participants | 30 [23.4 to 37.1] | 31 [25.7 to 37.3] | 14 [10.6 to 19.1]
Statistical Analysis 1: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants With an ISGA Score of 0 (Clear) or 1 (Almost Clear) at Weeks 1, 2, 4, 8, and 12
Description: Proportion of participants with at least a 2-Grade Improvement in ISGA was reported using a 5 point scale which indicates Score 0 (Clear): skin with no inflammatory or non-inflammatory lesions, Score 1 (Almost Clear): rare non-inflammatory lesions with no more than rare papules, Score 2 (Mild): greater than Grade 1, some non-inflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions), Score 3 (Moderate): greater than Grade 2, many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion, Score 4 (Severe): greater than Grade 3, many non-inflammatory and inflammatory lesions, but no more than a few nodular lesions and 5 (very severe): many non-inflammatory and inflammatory lesions and more than a few nodular lesions. May have cystic lesions. The investigator assessed ISGA score at baseline (Week 0/Day 1) and Weeks 1, 2, 4, 8, and 12. The area evaluated ISGA was limited to the face.
Time Frame: Week 1, 2, 4, 8, and 12
Population: ITT population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
Percentage of participants
  Week 1: number analyzed (Participants) | 200 | 287 | 295
  Week 1 | 2 [0.5 to 5.0] | 2 [0.8 to 4.5] | 1 [0.4 to 3.4]
  Week 2: number analyzed (Participants) | 197 | 281 | 297
  Week 2 | 7 [3.9 to 11.6] | 5 [2.5 to 7.8] | 5 [2.9 to 8.2]
  Week 4: number analyzed (Participants) | 191 | 269 | 296
  Week 4 | 11 [6.9 to 16.3] | 13 [9.2 to 17.6] | 7 [4.7 to 11.0]
  Week 8: number analyzed (Participants) | 186 | 260 | 292
  Week 8 | 22 [15.8 to 28.1] | 20 [15.3 to 25.4] | 9 [5.9 to 12.8]
  Week 12: number analyzed (Participants) | 184 | 262 | 290
  Week 12 | 30 [23.4 to 37.1] | 34 [27.9 to 39.7] | 20 [15.2 to 24.7]
Statistical Analysis 1: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 twice daily and CLDM twice daily at Week 1; Test type: Superiority or Other; p = 0.470, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 twice daily and CLDM twice daily at Week 2; Test type: Superiority or Other; p = 0.844, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 twice daily and CLDM twice daily at Week 4; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 twice daily and CLDM twice daily at Week 8; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 twice daily and CLDM twice daily at Week 12; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 once daily and CLDM twice daily at Week 1; Test type: Superiority or Other; p = 0.572, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 once daily and CLDM twice daily at Week 2; Test type: Superiority or Other; p = 0.335, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 once daily and CLDM twice daily at Week 4; Test type: Superiority or Other; p = 0.187, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 once daily and CLDM twice daily at Week 8; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of ISGA Score of 0 or 1 between GSK2585823 once daily and CLDM twice daily at Week 12; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Participants Who Have a Reduction of at Least 50 Percent in Total Lesions
Description: The percentage of participants who had reduction in total lesions (inflammatory and non-inflammatory) of at least 50 percent from Baseline at Weeks 1, 2, 4, 8, and 12 was measured.
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, and 12
Population: ITT population. Only those participants available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
Percentage of participants
  Week 1: number analyzed (Participants) | 200 | 287 | 295
  Week 1 | 18 [12.5 to 23.5] | 24 [19.5 to 29.8] | 15 [11.1 to 19.5]
  Week 2: number analyzed (Participants) | 201 | 289 | 299
  Week 2 | 47 [40.2 to 54.4] | 51 [44.9 to 56.8] | 32 [26.5 to 37.4]
  Week 4: number analyzed (Participants) | 201 | 289 | 299
  Week 4 | 63 [55.6 to 69.4] | 71 [65.3 to 76.1] | 52 [45.7 to 57.3]
  Week 8: number analyzed (Participants) | 201 | 289 | 299
  Week 8 | 79 [72.8 to 84.5] | 82 [77.1 to 86.3] | 69 [63.0 to 73.8]
  Week 12: number analyzed (Participants) | 201 | 289 | 299
  Week 12 | 85 [79.4 to 89.7] | 89 [84.3 to 92.0] | 79 [73.5 to 83.1]
Statistical Analysis 1: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of GSK2585823 twice daily and CLDM twice daily at Week 1; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of GSK2585823 twice daily and CLDM twice daily at Week 2; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of GSK2585823 twice daily and CLDM twice daily at Week 4; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of GSK2585823 twice daily and CLDM twice daily at Week 8; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: GSK2585823 Twice Daily vs CLDM Twice Daily; Comparison of GSK2585823 twice daily and CLDM twice daily at Week 12; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of GSK2585823 once daily and CLDM twice daily at Week 1; Test type: Superiority or Other; p = 0.480, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of GSK2585823 once daily and CLDM twice daily at Week 2; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of GSK2585823 once daily and CLDM twice daily at Week 4; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of GSK2585823 once daily and CLDM twice daily at Week 8; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: GSK2585823 Once Daily vs CLDM Twice Daily; Comparison of GSK2585823 once daily and CLDM twice daily at Week 12; Test type: Superiority or Other; p = 0.065, Cochran-Mantel-Haenszel

8. Secondary Outcome: Minimum Inhibitory Concentration (MIC) of Clinical Isolates to Antibiotics CLDM and Nadifloxacin (NDFX)
Description: MIC50 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 50% of isolates from a particular organism). MIC90 = minimum inhibitory concentration (minimum concentration of an agent that inhibits 90% of isolates from a particular organism) for the susceptibility of clinical isolates (Propionibacterium acnes before and after application of the CLDM and NDFX was reported. MIC50 and MIC90 values are single measurements for the entire population and not measured on a per-participant basis.
Time Frame: Baseline (Day 1) and Week12
Population: as for outcome 6
Measure: Number; unit: Micrograms/milliliter
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
Micrograms/milliliter
  CLDM,Baseline,MIC50: number analyzed (Participants) | 154 | 225 | 220
  CLDM,Baseline,MIC50 | 0.12 | 0.12 | 0.12
  CLDM,Baseline,MIC90: number analyzed (Participants) | 154 | 225 | 220
  CLDM,Baseline,MIC90 | 1 | 4 | 4
  CLDM, Week 12,MIC50: number analyzed (Participants) | 12 | 22 | 59
  CLDM, Week 12,MIC50 | 0.25 | 0.5 | 0.5
  CLDM, Week 12,MIC90: number analyzed (Participants) | 12 | 22 | 59
  CLDM, Week 12,MIC90 | 128 | 128 | 128
  NDFX,Baseline,MIC50: number analyzed (Participants) | 154 | 225 | 220
  NDFX,Baseline,MIC50 | 0.25 | 0.25 | 0.25
  NDFX,Baseline,MIC90: number analyzed (Participants) | 154 | 225 | 220
  NDFX,Baseline,MIC90 | 0.5 | 0.5 | 0.5
  NDFX, Week 12,MIC50: number analyzed (Participants) | 12 | 22 | 59
  NDFX, Week 12,MIC50 | 0.25 | 0.25 | 0.25
  NDFX, Week 12,MIC90: number analyzed (Participants) | 12 | 22 | 59
  NDFX, Week 12,MIC90 | 0.5 | 0.5 | 0.5

9. Secondary Outcome: Change in Investigator Assessment of Tolerability (Erythema, Dryness and Peeling) From Baseline to Weeks 1, 2, 4 and 8 and 12
Description: Erythema (redness), dryness, and peeling, were evaluated independently by the investigator on a five point scale from 0 to 4 defined as 0-none, 1-very minimal, 2-mild, 3-moderate, 4-severe. Day 1 was Baseline and Change from Baseline was calculated by subtracting Baseline value from value at specified time points (Week 1, 2, 4, 8, and 12).
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8, and 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
Score on scale
  Erythema score-Week 1: number analyzed (Participants) | 198 | 285 | 298
  Erythema score-Week 1 | -0.11 (0.58) | -0.00 (0.63) | -0.11 (0.52)
  Erythema score-Week 2: number analyzed (Participants) | 192 | 275 | 297
  Erythema score-Week 2 | -0.16 (0.76) | -0.02 (0.82) | -0.19 (0.58)
  Erythema score-Week 4: number analyzed (Participants) | 187 | 266 | 294
  Erythema score-Week 4 | -0.30 (0.72) | -0.24 (0.75) | -0.27 (0.62)
  Erythema score-Week 8: number analyzed (Participants) | 185 | 262 | 291
  Erythema score-Week 8 | -0.43 (0.82) | -0.33 (0.78) | -0.31 (0.67)
  Erythema score-Week 12: number analyzed (Participants) | 183 | 262 | 290
  Erythema score-Week 12 | -0.49 (0.82) | -0.45 (0.87) | -0.38 (0.75)
  Dryness yscore-Week 1: number analyzed (Participants) | 198 | 285 | 298
  Dryness yscore-Week 1 | 0.10 (0.65) | 0.29 (0.76) | -0.04 (0.47)
  Dryness score-Week 2: number analyzed (Participants) | 192 | 275 | 297
  Dryness score-Week 2 | 0.04 (0.65) | 0.23 (0.80) | -0.11 (0.51)
  Dryness score-Week 4: number analyzed (Participants) | 187 | 266 | 294
  Dryness score-Week 4 | -0.06 (0.57) | 0.00 (0.65) | -0.15 (0.53)
  Dryness score-Week 8: number analyzed (Participants) | 185 | 262 | 291
  Dryness score-Week 8 | -0.11 (0.61) | -0.00 (0.67) | -0.13 (0.50)
  Dryness score-Week 12: number analyzed (Participants) | 183 | 262 | 290
  Dryness score-Week 12 | -0.18 (0.62) | -0.10 (0.61) | -0.17 (0.52)
  Peeling score-Week 1: number analyzed (Participants) | 198 | 285 | 298
  Peeling score-Week 1 | 0.09 (0.50) | 0.19 (0.68) | -0.04 (0.39)
  Peeling score-Week 2: number analyzed (Participants) | 192 | 275 | 297
  Peeling score-Week 2 | 0.02 (0.49) | 0.17 (0.68) | -0.10 (0.39)
  Peeling score-Week 4: number analyzed (Participants) | 187 | 266 | 294
  Peeling score-Week 4 | -0.05 (0.44) | 0.04 (0.54) | -0.14 (0.43)
  Peeling score-Week 8: number analyzed (Participants) | 185 | 262 | 291
  Peeling score-Week 8 | -0.08 (0.46) | 0.03 (0.56) | -0.13 (0.43)
  Peeling score-Week 12: number analyzed (Participants) | 183 | 262 | 290
  Peeling score-Week 12 | -0.08 (0.49) | -0.07 (0.51) | -0.13 (0.44)

10. Secondary Outcome: Change in Participant Assessment of Tolerability ( Itching and Burning/Stinging ) From Baseline to Weeks 1, 2, 4, 8 and 12
Description: Burning/stinging, itching were evaluated independently by the participant on a five point scale from 0 to 4 defined as 0-none, 1-very minimal, 2-mild, 3-moderate, 4-severe. Day 1 was Baseline and Change from Baseline was calculated by subtracting Baseline value from value at specified time points (Week 1, 2, 4, 8, and 12).
Time Frame: Baseline (Day 1) and Week 1, 2, 4, 8 and 12
Population: ITT population. Only those participants available at the specified time points were analyzed (represented by n=X. X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
Number analyzed (Participants) | 204 | 296 | 299
Score on scale
  Itching Score, Week 1: number analyzed (Participants) | 198 | 285 | 298
  Itching Score, Week 1 | -0.02 (0.53) | 0.07 (0.61) | -0.08 (0.53)
  Itching Score, Week 2: number analyzed (Participants) | 192 | 275 | 297
  Itching Score, Week 2 | -0.06 (0.58) | 0.12 (0.73) | -0.13 (0.48)
  Itching Score, Week 4: number analyzed (Participants) | 187 | 266 | 294
  Itching Score, Week 4 | -0.10 (0.51) | -0.02 (0.48) | -0.14 (0.51)
  Itching Score, Week 8: number analyzed (Participants) | 185 | 262 | 291
  Itching Score, Week 8 | -0.15 (0.50) | -0.06 (0.43) | -0.14 (0.55)
  Itching Score, Week 12: number analyzed (Participants) | 183 | 262 | 290
  Itching Score, Week 12 | -0.10 (0.59) | -0.08 (0.53) | -0.12 (0.52)
  Burning/Stinging Score, Week 1: number analyzed (Participants) | 198 | 285 | 298
  Burning/Stinging Score, Week 1 | 0.08 (0.55) | 0.26 (0.76) | -0.02 (0.45)
  Burning/Stinging Score, Week 2: number analyzed (Participants) | 192 | 275 | 297
  Burning/Stinging Score, Week 2 | 0.02 (0.45) | 0.11 (0.61) | -0.06 (0.37)
  Burning/Stinging Score, Week 4: number analyzed (Participants) | 187 | 266 | 294
  Burning/Stinging Score, Week 4 | -0.02 (0.43) | -0.02 (0.48) | -0.07 (0.39)
  Burning/Stinging Score, Week 8: number analyzed (Participants) | 185 | 262 | 291
  Burning/Stinging Score, Week 8 | -0.02 (0.44) | -0.04 (0.47) | -0.08 (0.39)
  Burning/Stinging Score, Week 12: number analyzed (Participants) | 183 | 262 | 290
  Burning/Stinging Score, Week 12 | -0.06 (0.38) | -0.08 (0.38) | -0.08 (0.37)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 throughout the treatment period up to Week 12. There were no serious adverse events in this study. Data has been presented for non serious adverse events up to Week 12.
Description: ITT population was used.
Arm/Group | GSK2585823 Once Daily | GSK2585823 Twice Daily | CLDM Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/296 | 0/299
Serious Adverse Events (participants affected / at risk) | 0/204 | 0/296 | 0/299
Other Adverse Events (participants affected / at risk) | 108/204 | 163/296 | 110/299
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2585823 Once Daily (N=204) | GSK2585823 Twice Daily (N=296) | CLDM Twice Daily (N=299)
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 35 | 8
Dermatitis contact (Skin and subcutaneous tissue disorders) | 14 | 24 | 5
Erythema (Skin and subcutaneous tissue disorders) | 8 | 22 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 17 | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 25 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 10 | 7
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 4 | 6 | 4
Skin irritation (Skin and subcutaneous tissue disorders) | 3 | 8 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 4 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 28 | 48 | 39
Influenza (Infections and infestations) | 4 | 9 | 7
Gastroenteritis (Infections and infestations) | 3 | 2 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 2 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Infected dermal cyst (Infections and infestations) | 2 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0
Pericoronitis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 4
Blood bilirubin increased (Investigations) | 1 | 2 | 5
White blood cell count increased (Investigations) | 1 | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 4
Glucose urine present (Investigations) | 1 | 1 | 2
Protein urine present (Investigations) | 2 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 6 | 12 | 4
Headache (Nervous system disorders) | 2 | 3 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Facial pain (General disorders) | 9 | 9 | 4
Pyrexia (General disorders) | 2 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0
Nodule (General disorders) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Radicular cyst (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 2 | 2 | 0
Erythema of eyelid (Eye disorders) | 1 | 2 | 0
Blepharitis (Eye disorders) | 1 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Eyelid irritation (Eye disorders) | 0 | 2 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Eczema eyelids (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0
Eyelids pruritus (Eye disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.